CLINICAL TRIAL: NCT02668133
Title: Efficacy of Exogenous Phytase Added to Small Quantity Lipid Nutrient Supplements (SQ-LNS) on the Fractional and Total Absorption of Zinc Among Young Children in the Gambia: A Double-blind Randomized Controlled Trial With a Cross-over Design
Brief Title: Zinc Absorption From SQ-LNS With and Without Phytase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: SCC 1420
Record Dates: First submitted 2016-01-21; First posted 2016-01-29 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Individuals at Risk of Zinc Deficiency
Keywords: zinc deficiency; zinc absorption

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lipid-based nutrient supplement SQ-LNS (Active Comparator): • Small quantity lipid nutrient supplement SQ-LNS containing 6 mg iron and 8 mg zinc per 20 g sachet (per day) 0.9 mg isotopically enriched 67Zn,0.30 mg isotopically enriched 70Zn, 0.60 mg non-enriched zinc delivered orally in sugar solution
  1 mg isotopically enriched 68Zn intravenously
  Interventions: Dietary Supplement: the nutritional supplement to be used in this trial is a SQ-LNS; Dietary Supplement: 0.9 mg isotopically enriched 67Zn,0.30 mg isotopically enriched 70Zn, 0.60 mg non-enriched zinc; Dietary Supplement: 1 mg isotopically enriched 68Zn
- lipid-based nutrient supplement SQ-LNS with phytase (Experimental): • Small quantity lipid nutrient supplement SQ-LNS containing 6 mg iron and 8 mg zinc per 20 g sachet (per day). Exogenous phytase (projected concentration ~500 FTU/20 g SQ-LNS added during manufacturing 0.9 mg isotopically enriched 67Zn,0.30 mg isotopically enriched 70Zn, 0.60 mg non-enriched zinc delivered orally in sugar solution
  1 mg isotopically enriched 68Zn intravenously
  Interventions: Dietary Supplement: lipid-based nutrient supplement (SQ-LNS) with phytase; Dietary Supplement: 0.9 mg isotopically enriched 67Zn,0.30 mg isotopically enriched 70Zn, 0.60 mg non-enriched zinc; Dietary Supplement: 1 mg isotopically enriched 68Zn

INTERVENTIONS:
Dietary Supplement: the nutritional supplement to be used in this trial is a SQ-LNS — Small quantity lipid nutrient supplement (SQ-LNS) containing 6 mg iron and 8 mg zinc per 20 g sachet (per day
  Arms: lipid-based nutrient supplement SQ-LNS
Dietary Supplement: lipid-based nutrient supplement (SQ-LNS) with phytase — • Small quantity lipid nutrient supplement (SQ-LNS) containing 6 mg iron and 8 mg zinc per 20 g sachet (per day). Exogenous phytase (projected concentration ~500 FTU/20 g SQ-LNS) added during manufacturing
  Arms: lipid-based nutrient supplement SQ-LNS with phytase
Dietary Supplement: 0.9 mg isotopically enriched 67Zn,0.30 mg isotopically enriched 70Zn, 0.60 mg non-enriched zinc — delivered orally in sugar solution
Dietary Supplement: 1 mg isotopically enriched 68Zn — administered intravenously

SUMMARY:
Background: Community based-intervention trials conducted among infants and young children in low- and middle-income countries have found that zinc supplementation of young children (in the form of liquid supplements or dispersible tablets) increases linear growth and weight gain, and reduces the prevalence of diarrhea and respiratory infections, and lowers all-cause mortality. Aside from supplements, additional dietary zinc can also be provided through "home-fortification" of complementary foods with small-quantity lipid-based nutrient supplements (SQ-LNS; 20g/d), which are typically formulated as a peanut-based paste enriched with a vitamin and mineral complex containing 8 mg elemental zinc (as ZnSO4). However, the efficacy of LNS as a delivery vehicle for preventive zinc supplementation remains uncertain. Two recent studies, which provided LNS containing 4-10 mg Zn daily for 6-9 months found no significant differences in plasma zinc concentrations at the end of the intervention period compared to placebo.

This lack of response may be due to the reduced absorption of zinc when it is part of a complex food matrix and provided with cereal-based meals; both SQ-LNS and cereal grains contain moderate to high concentrations of phytate, the main dietary factor known to substantially reduce zinc absorption. The addition of exogenous phytases is an efficacious strategy to reduce the phytate content of foods, and increase the bioavailability of dietary zinc; however, the efficacy of this approach has not yet been demonstrated for SQ-LNS.

Objective: The overall objective of the study is to assess the efficacy of adding exogenous phytase to SQ-LNS by investigating intra-individual differences in the fractional absorption of zinc (FAZ) among children who receive additional dietary zinc (8 mg/d) from SQ-LNS with or without phytase.

Trial approach: The study will be a double-blind randomized controlled clinical trial, designed to permit within-child comparisons of zinc absorption from SQ-LNS, with or without exogenous phytase, by using the triple stable-isotope ratio tracer technique. The clinical study will enroll 34 children between the ages of 18-23 months. The main outcome of interest is the intra-individual difference in the FAZ from porridge-based meals containing SQ-LNS with and without phytase. Up to an' additional 36 children will be enrolled in a pilot feeding study to determine portion sizes of study meals.

Trial setting: Keneba, The Gambia

Trial interventions:

The SQ-LNS (20g) used in this study will be provided by Nutriset, S.A.S. The exogenous phytase (DSM phytase Tolerase 20000G) is derived from Aspergillus niger; phytase will be added to the SQ-LNS during the production phase, and will be enzymatically active in vivo at the time of consumption.

Feeding Protocol and Study Diet: The study diet for the 2day absorption study will consist of the following: 1) Two stable-isotope labeled test meals per day (porridge made from locally procured non-fermented cereal, mixed with 10 g of SQ-LNS), with children randomized to receive either SQ-LNS with phytase or SQ-LNS without phytase on the first day and the alternative product on the second; 2) One additional standardized meal per day (e.g. rice with sauce); 3) Low-zinc, low-phytate food (e.g. bananas) consumed ad libitum if requested (with the exception of 1 hour before and 2 hours after each test meal). Children will be fed by their caregivers under supervision by a study fieldworker. The SQ-LNS product (without phytase) will be provided to children twice per day for one day prior to the start of the stable isotope absorption studies, in order to habituate children to the study diet and location. Children will attend the study clinic daily for four days and will be enrolled in the study for a total of ten days.

Zinc absorption studies: The FAZ of zinc will be measured by a triple-isotope tracer ratio technique, using orally administered extrinsic labels (Zn-67 and Zn-70) and intravenous Zn-68. Urine samples, collected pre- and post-isotope administration (d 1, 5-9) will be analyzed for zinc isotope ratios by ICP-MS. FAZ will be calculated based on the mean isotopic ratios obtained from the enriched urine samples, and based on the tracer:tracee ratio method. TAZ will be calculated by multiplying FAZ by total zinc intake from the test meals.

Data Collection: The following information will be collected from each subject: brief medical history; physical examination; weight and height; daily morbidity and pre-intervention blood sampling for hemoglobin, complete blood count and plasma zinc concentration, malaria and systemic inflammation (C-reactive protein and α-1-acid glycoprotein).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from at least one parent, including consent for samples to be shipped outside of The Gambia
* Age 18-23 months
* non-breast feeding children and consumption of coos porridge
* Previous consumption of peanut based products with no known adverse reaction

Exclusion Criteria:

* Weight-for-height z-score (WHZ) <-3 Z with respect to WHO 2006 standards*
* Presence of bipedal oedema
* Severe illness warranting hospital referral
* Congenital abnormalities potentially interfering with micronutrient metabolism
* Chronic medical condition (e.g. malignancy) requiring frequent medical attention
* Known HIV infection of index child or child's mother
* Currently consuming vitamin or mineral supplements or zinc- or iron-fortified infant formulas/foods
* Diarrhoea (>3 liquid or semi-liquid stools per day) within the past 7 days
* Symptomatic acute or chronic febrile infection within the past 7 days
* Hemoglobin < 70 g/L*
* Positive rapid diagnostic test for malaria antigenemia (HRP2)* * Exclusion criteria for main metabolic study only (not criteria for the pilot feeding study, as anthropometric and biochemical data will not be collected

Ages: 18 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
Fractional absorption of zinc | 10 days
  Fractional absorption of zinc is estimated using the triple zinc stable isotope tracer ratio technique. 67Zn and 70Zn are administered orally and 68Zn is administered intravenously. The urinary enrichment of the three isotopes is measured over 5 days (ICP-MS) and tracer:tracee ratios are calculated.

SECONDARY OUTCOMES:
Total absorption of zinc | 10 days
  Total absorption of zinc is estimated by multiplying fractional absorption of zinc by dietary zinc intake.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Prentice, PhD, Principal Investigator — Medical Research Council The Gambia
Locations (1):
- Keneba Clinic, Kiang, The Gambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zyba SJ, Wegmuller R, Woodhouse LR, Ceesay K, Prentice AM, Brown KH, Wessells KR. Effect of exogenous phytase added to small-quantity lipid-based nutrient supplements (SQ-LNS) on the fractional and total absorption of zinc from a millet-based porridge consumed with SQ-LNS in young Gambian children: a randomized controlled trial. Am J Clin Nutr. 2019 Dec 1;110(6):1465-1475. doi: 10.1093/ajcn/nqz205. PMID 31504101